CLINICAL TRIAL: NCT01257776
Title: Using Mesenchymal Stem Cells From Adipose Tissue (CeTMAd) as Cell Regeneration Therapy in Chronic Ischemic Syndrome of Lower Limbs in Diabetic Patients
Brief Title: Human Adipose Derived Mesenchymal Stem Cells for Critical Limb Ischemia (CLI) in Diabetic Patients
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Andalusian Initiative for Advanced Therapies - Fundación Pública Andaluza Progreso y Salud (Other)
Collaborators: Iniciativa Andaluza en Terapias Avanzadas (Other)
Responsible Party: Sponsor
Organization: Andalusian Network for Design and Translation of Advanced Therapies (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CeTMAd/ICPD/2008; NCT01079403 (obsolete NCT alias)
Record Dates: First submitted 2010-12-09; First posted 2010-12-10 (Estimated); Last update posted 2015-08-05 (Estimated); Status verified 2014-11

CONDITIONS: Critical Limb Ischemia (CLI); Diabetes
Keywords: Critical Limb Ischemia (CLI); Diabetes; Mesenchymal Stem Cells; Regenerative Therapy
MeSH Terms: conditions — Chronic Limb-Threatening Ischemia; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Mesenchymal stem cells 0,5 million * weight (kg) (Active Comparator): Group of low dose of Mesenchymal stem cells.
  Interventions: Drug: Autologous adipose derived mesenchymal stem cells
- Mesenchymal stem cells 1 million * weight (kg) (Active Comparator): Group of mid dose of mesenchymal stem cells
  Interventions: Drug: Autologous adipose derived mesenchymal stem cells
- Controlled group (No Intervention): Controlled group with no intervention

INTERVENTIONS:
Drug: Autologous adipose derived mesenchymal stem cells — Intra-arterial administration through a selective cannulation of target common femoral artery
  Arms: Mesenchymal stem cells 0,5 million * weight (kg); Mesenchymal stem cells 1 million * weight (kg)

SUMMARY:
A prospective, multicenter, open, randomized, parallel-group controlled study for two levels of dose.

The study population will consist of 30 non-diabetic patients with critical chronic ischemia in at least one of the lower limbs (CLI) and without possibility of revascularization, from whom results can clinically be evaluable, of whom, 20 patients will be included in the experimental group (10 for each dose level) and 10 in the control group.

In each of the two dose levels to be used in the study, 15 patients will be included, who will be randomized to the experimental group or the control group according to a distribution 2:1 (2 patients in the experimental group and 1 in control group), thus at each dose level, we will have 10 patients in the experimental group (treated with mesenchymal cells of adipose tissue) and 5 patients in the control group (conventional treatment)

ELIGIBILITY:
Inclusion Criteria:

* Diabetes, type 1 or 2
* Critical Limb Ischemia (Rutherford Becker Class II,III or IV)of at least one limb.
* No options for target limb revascularization.

Exclusion Criteria:

* Cancer antecedent in the last two years
* Current limb infection or limb gangrene

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2010-12; Primary Completion 2013-02 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Angiographic assessment of neovasculogenesis (angiogenesis plus arteriogenesis) | 6 months
  Target limb vascularization would be quantified by a dedicated software, MetaMorph® v.6.3, by using Angiogenesis Tube Formation application module. Neovasculogenesis would be the difference between vascularization at baseline and 6 months follow-up.
Major adverse event (death, target limb amputation) | 1 month, 6 months, 12 months

SECONDARY OUTCOMES:
Ankle Brachial Index | 1 month, 6 months, 12 months
University of Texas Classification at target limb | 1 month, 6 months, 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Rafael J Ruiz-Salmeron, MD, PhD, Principal Investigator — University Hospital Virgen Macarena. Seville.Spain; Antonio De la Cuesta, MD, Principal Investigator — University Hospital Virgen Macarena. Seville.Spain
Locations (2):
- Spain (2):
  - University Hospital Virgen Macarena, Seville, Seville
  - CABIMER (Andalusian Center for Molecular Biology and Regenerative Medicine), Seville, Seville